CLINICAL TRIAL: NCT01815541
Title: Administration of Subcutaneous Teicoplanin in the Treatment of Osteoarticular Infections: Tolerance Study
Acronym: TEICOPLANIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2012_843_0008; 2012-003690-25 (EudraCT Number)
Record Dates: First submitted 2013-03-15; First posted 2013-03-21 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Osteoarticular Infection
Keywords: subcutaneous teicoplanin; osteoarticular; infections; tolerance; teicoplanin
MeSH Terms: conditions — Infections | interventions — Teicoplanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- teicoplanin (Experimental): this group receive the teicoplanin
  Interventions: Drug: teicoplanin

INTERVENTIONS:
Drug: teicoplanin

SUMMARY:
This is a biomedical research, prospective, mono centric, tolerance study Of the administration of subcutaneous teicoplanin in the treatment of osteoarticular infections.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Inpatient orthopedic surgery
* Achieved a bone and joint infection documented gram + (staphylococci golden coagulase-negative staphylococci, enterococci, streptococci)
* Bacteria resistant to lincosamides, quinolones and rifampicin
* Bacteria susceptible to teicoplanin (MIC ≤ 4 mg / L)
* Balanced patient teicoplanin administered intravenously (2 successive doses between 30 and 40 mg / mL)

Exclusion Criteria:

* Patient not affiliated to the social security
* Pregnant and lactating women
* Known hypersensitivity to teicoplanin (rash, ...)
* Patients with a central catheter or an implantable chamber
* Patient hemodialysis
* Patient has another participant biomedical research on a drug to prevent drug interactions
* Patient minor
* Patient major protected (protection of the court, wardship, trusteeship)
* Patient admitted for emergency or incapable of consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
measure of tolerance | 6 weeks
  The frequencies of adverse reactions at the injection site SC will be measured to assess the local tolerance of teicoplanin by SC.

CONTACTS AND LOCATIONS:
Overall Officials: Youssef El SAMAD, PH, Principal Investigator — CHU Amiens, France
Locations (1):
- CHU Amiens, Amiens, Picardie, France

REFERENCES:
- [Result] El Samad Y, Lanoix JP, Bennis Y, Diouf M, Saroufim C, Brunschweiler B, Rousseau F, Joseph C, Hamdad F, Ait Amer Meziane M, Routier S, Schmit JL. Tolerability and Plasma Drug Level Monitoring of Prolonged Subcutaneous Teicoplanin Treatment for Bone and Joint Infections. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6365-8. doi: 10.1128/AAC.00351-16. Print 2016 Oct. PMID 27458228